CLINICAL TRIAL: NCT07245836
Title: Anti-inflammatory Effects and Clinical Efficacy of Topical Thealoz Total Eye Drops in Patients With Chronic Dry Eye Disease and Associated Ocular Surface Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc. Prof. Priv. Doz. Dr., PhD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2769-005
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry eye disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thealoz Total® eye drops (Experimental): Thealoz Total® eye drops; 3-6 Drops per day for 12 weeks
  Interventions: Drug: Thealoz Total® Eye Drops, Laboratoires Thea, Clermont Ferrand, France

INTERVENTIONS:
Drug: Thealoz Total® Eye Drops, Laboratoires Thea, Clermont Ferrand, France — topical lubrication

SUMMARY:
Dry eye disease (DED) is a highly prevalent ocular condition and induces a significant burden to the affected patients. Regardless of the underlying etiology, DED is associated with increased inflammation of the entire ocular surface including the adnexa, conjunctiva and cornea. As such, there is evidence from in vitro, animal and clinical studies that this inflammatory response of the ocular surface plays a pathophysiological key role in the development of DED. The Dry Eye Workshop 2007 (DEWS) therefore suggests beside of restoring the tear film by administering topical lubricants, breaking the vicious circle of inflammation is an important mainstay of therapy in patients with DED. Recently, a new medical device (Thealoz Total® eye drops) has been introduced for the treatment DED. Thealoz Total® eye drops are based on hyaluronic acid and exert their main action by lubricating the ocular surface. Further, this new formulation offers several advantages that make them potentially interesting to reduce DED related symptoms. First, the formulation is preservative-free, which is of special importance in patients with DED, since it has been shown that preservatives are detrimental for the ocular surface. thereby reducing signs and symptoms related to DED. Secondly, in addition to the lubricating effect of hyaluronic acid, Thealoz Total eye drops also contain trehalose, which exerts osmoprotetive effects and N-Acetyl Aspartyl Glutamic Acid (NAAGA). NAAGA is an amino conjugated dipeptide with anti-inflammatory properties. Thus, it is reasonable to hypothesize that Thealoz total eye drops are also capable of reducing ocular surface inflammation. The aim of the present study is to investigate whether topical administration with Thealoz Total® improves ocular surface inflammation as well as clinical signs and symptoms associated with DED.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Normal ophthalmic findings except dry eye disease
* Chronic dry eye defined as longer than six months since diagnosis
* OSDI ≥ 22
* Conjunctival Hyperemia≥ Grade 3 (Efron Scale)
* Current use of topical lubricants since at least 3 months

Exclusion Criteria:

Ophthalmic exclusion criteria

- Best far corrected visual acuity < 1/10

Severe Dry Eye associated with:

* Eyelid malposition
* Stevens Johnson Syndrome
* Corneal dystrophy
* Ocular neoplasia
* Filamentous keratitis
* Corneal neovascularisation
* Orbital radiotherapy
* Dry eye related to GVHD

History of any of the following within last 3 months:

* Systemic treatment of dry eye
* Systemic treatment of MGD
* Isotretinoïde,
* Cyclosporine,
* Tacrolimus, Siromilus, Pimecrolimus
* Punctual plugs

History of any of the following within previous six months:

* ocular trauma
* ocular infection, Ocular allergy

History of any of the following within last 12 months:

* inflammatory corneal ulcer
* Herpetic eye infection or uveitis
* Ocular surgery

Systemic / non ophthalmic exclusion criteria:

- Known hypersensitivity to any of the components of the medical device under investigation or other study medication

Specific exclusion criteria for women:

* Pregnant or breast-feeding woman.
* Woman of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (i.e. hormonal contraceptives, intra-uterine device, contraceptive implant or condoms)

Exclusion criteria related to general conditions

- Inability of patient to understand the investigation procedures and thus inability to give valid, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-07-06 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction assessed by a VAS | week 12
  Patient satisfaction assessed by a Visual Analogue Scale (VAS) (min 0 - max 100)
  The VAS consists of a 10cm line, with two end points representing 0 ('no symptoms') and 100 ('max symptoms')
Conjunctival hyperemia grading with Photographs (Efron) scale at week 12 | week 12
  Conjunctival hyperemia grading with Photographs (Efron) scale at week 12
  The Efron Scale is a clinical grading scale used to assess conjunctival hyperemia.
  It provides a standardized visual grading from 0 to 4 Grade 0 = normal Grade 1 = trace / very mild Grade 2 = mild to moderate Grade 3 = moderate to severe Grade 4 = severe

SECONDARY OUTCOMES:
Changes from baseline in conjunctival hyperemia grading with photographs (Efron) scale | week 6 and 12
  Changes from baseline in conjunctival hyperemia grading with photographs (Efron) scale
  The Efron Scale is a clinical grading scale used to assess conjunctival hyperemia.
  It provides a standardized visual grading from 0 to 4 Grade 0 = normal Grade 1 = trace / very mild Grade 2 = mild to moderate Grade 3 = moderate to severe Grade 4 = severe
Changes from baseline in corneal fluorescein staining according to the Oxford Scale | week 6 and 12
  Changes from baseline in corneal fluorescein staining according to the Oxford Scale
  The Oxford Scale is a standardized grading system corneal staining after fluorescein dye application. It indicates the level of epithelial damage or ocular surface compromise.
  The grading runs from 0 to 5, based on a set of reference panels with dots representing staining patterns.
  Grade 0 = none (no staining) Grade 1 = trace (minimal staining, very few punctate dots) Grade 2 = mild (slightly more numerous dots) Grade 3 = moderate (obvious punctate staining, more confluent areas) Grade 4 = marked (extensive staining, coalescent areas) Grade 5 = severe (dense, widespread staining, severe epithelial damage)
Changes from baseline in Tear Break Up Time (BUT) with Minims- Fluorescein Sodium 2,0% | week 6 and 12
  Changes from baseline in Tear Break Up Time (BUT) with Minims- Fluorescein Sodium 2,0%
Changes from baseline in Schirmer I test using Schirmer paper strips | week 6 and 12
  Changes from baseline in Schirmer I test using Schirmer paper strips
Changes from baseline in conjunctival hyperaemia assessment using Mc Monnies photographic scale | week 6 and 12
  Changes from baseline in conjunctival hyperaemia assessment using Mc Monnies photographic scale
  The McMonnies Photographic Scale is a clinical grading system for bulbar conjunctival hyperemia.
  It uses a series of standardized photographs of eyes with increasing levels of redness.
  Clinicians compare the patient's eye to these photographs and assign a grade.
  The scale typically ranges from 0 to 5:
  0 = none (normal, no redness)
  1. = trace (very mild hyperemia)
  2. = mild
  3. = moderate
  4. = marked
  5. = severe (intense hyperemia with engorged vessels)
Changes from baseline in symptoms using the OSDI questionnaire | week 6 and 12
  Changes from baseline in symptoms using the Ocular Surface Disease Index (OSDI) questionnaire
  It contains 12 questions, divided into three domains, every qestion has 0-4 points:
  * Ocular symptoms
  * Vision-related function
  * Environmental triggers
  Interpretation of scores:
  0-12 = normal 13-22 = mild dry eye 23-32 = moderate dry eye 33-100 = severe dry eye
  Not every patient will necessarily answer all 12 questions. To account for this, the OSDI uses a normalization formula:
  1. Add together all the scores from the answered questions.
  2. Multiply this sum by 25 (this scales the score to a 0-100 range).
  3. Divide the result by the number of questions answered.
Changes from baseline in symptoms within the last 48 hours | week 6 and 12
  Changes from baseline in symptoms within the last 48 hours
  Patient will be asked: "How do you judge the severity of your following ocular symptoms within the last 48 hours?"
  The severity of the following ocular symptoms will be assessed at each visit: burning/irritation, stinging/eye pain, light sensitivity, itching/pruritus, eye dryness feeling, tearing, foreign body sensation as follows:
  0 = Absent
  1. = Mild, present but not disturbing
  2. = Moderate, disturbing, but not limiting with daily activities
  3. = Severe, very distressing and interfering with daily activities The ocular symptoms will be assessed in global for both eyes at each visit. The value at Visit 1 will be the baseline value.
  Questions are:
  Burning/irritation Burning/pain Light sensitivity (photophobia) Itching Sensation of dryness in the eyes Tearing (watery eyes) Foreign body sensation
Changes from baseline in tear proteomics and lipidomics | week 12
  Changes from baseline in tear proteomics and lipidomics
  Tear film samples will be collected on week 1 and week 12 by Schirmer-I-Test. Samples will be extracted and and measured in an untargeted fashion.
  Samples will be stored at -80°C until time of analysis and will be discarded after analysis.
Patient satisfaction assessed by a VAS | week 12
  Patient satisfaction assessed by a Visual Analogue Scale (VAS)
  The VAS consists of a 10cm line, with two end points representing 0 ('minimum') and 100 ('maximum')

OTHER OUTCOMES:
Adverse events | Week 0 - 12
  Adverse events
Best corrected distance visual acuity. | Week 0 - 12
  Best corrected distance visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No